CLINICAL TRIAL: NCT07195214
Title: Effect of Dexmedetomidine on Recurrent Laryngeal Nerve Monitoring: A Prospective Observational Comparative Study With Midazolam
Brief Title: EFFECT OF DEXMEDETOMİDİNE ON RECURRENT LARYNGEAL NERVE MONİTORİNG: A COMPARATİVE STUDY WİTH MİDAZOLAM
Acronym: DEX-RLN
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Other Study IDs: Se; E-30640013-050.04-246788 (Other: Amasya University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Surgery Intraoperative Nerve Monitoring (IONM) Recurrent Laryngeal Nerve Function Dexmedetomidine vs Midazolam (Anesthetic Agents)
Keywords: Thyroid surgery; intraoperative neuromonitoring (IONM); total intravenous anesthesia; dexmedetomidine; midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dexmedetotimidine: using dexmedetotimidine
- midazolam: uzing midazolam

SUMMARY:
This prospective observational study evaluated the effect of dexmedetomidine compared with midazolam on intraoperative monitoring of the recurrent laryngeal nerve during thyroid surgery. The main goal was to assess whether dexmedetomidine influences the time to identify the recurrent laryngeal nerve and the quality of nerve signals. Secondary outcomes included time to vagus nerve identification, intraoperative hemodynamic changes, extubation time, postoperative nausea and vomiting, sedation levels, and recovery parameters. A total of 60 adult patients undergoing thyroidectomy with intraoperative neuromonitoring were included. The findings are expected to guide anesthetic choices that optimize patient safety and surgical outcomes in thyroid operations.

DETAILED DESCRIPTION:
This prospective observational study was conducted to investigate the effect of dexmedetomidine compared with midazolam on intraoperative monitoring of the recurrent laryngeal nerve (RLN) during thyroid surgery. Sixty adult patients scheduled for thyroidectomy under general anesthesia with intraoperative nerve monitoring were enrolled. Patients were allocated to receive either dexmedetomidine or midazolam as part of anesthesia induction. The primary objective was to compare the time required to identify the recurrent laryngeal nerve and the quality of electromyographic signals between the two groups. Secondary outcomes included time to vagus nerve identification, intraoperative hemodynamic changes such as bradycardia or hypotension, amplitude and latency of RLN signals, extubation time, postoperative nausea and vomiting, sedation scores, and length of stay in the post-anesthesia care unit. The study was approved by the Amasya University Non-Interventional Clinical Research Ethics Committee (Approval No: E-30640013-050.04-246788). Findings from this study may contribute to optimizing anesthetic protocols for thyroid surgery to improve patient safety and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years Patients scheduled for elective thyroidectomy under general anesthesia American Society of Anesthesiologists (ASA) physical status I-II Planned use of intraoperative nerve monitoring (IONM) Provided written informed consent

Exclusion Criteria:

Previous neck surgery or radiotherapy affecting recurrent laryngeal nerve anatomy Pre-existing vocal cord paralysis or laryngeal nerve dysfunction Severe cardiovascular disease (e.g., advanced heart block, uncontrolled hypertension) Severe hepatic or renal dysfunction Known allergy or contraindication to dexmedetomidine, midazolam, or study medications Pregnancy or breastfeeding Refusal to participate or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients (aged 18-65 years) scheduled for elective thyroidectomy under general anesthesia with intraoperative nerve monitoring. All participants were ASA physical status I-II, had no pre-existing laryngeal nerve dysfunction, and provided written informed consent. Patients were recruited at Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, Department of General Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Time to Identification of the Recurrent Laryngeal Nerve (minutes) | Intraoperative period (from skin incision until RLN identification, typically within the first 60 minutes of surgery).
  The interval between the start of intraoperative neuromonitoring and the successful identification of the recurrent laryngeal nerve during thyroidectomy. This measure evaluates whether dexmedetomidine or midazolam affects the speed of RLN identification.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya Univessity, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of ethical considerations and local regulations. Only summarized and de-identified results will be published in scientific journals.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT07195214/ICF_000.pdf